CLINICAL TRIAL: NCT07112027
Title: Exploration of the Neural Correlates of Social Expertise: an Fmri Study Comparing Healthy Individuals With Different Levels and Types of Expertise
Brief Title: Exploring the Relationship Between Social Expertise and Ability to Process Different Types of Abstract Concepts and the Neural Resources Allocated to Their Processing
Acronym: EXPERTISE-SOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Jubin Abutalebi, Director Center for Neurolinguistics and Psycholinguistics (CNPL), Università Vita-Salute San Raffaele
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: EXPERTISE-SOC; 2022YJA4TB (Other Grant/Funding Number: Ministero dell'Università e della Ricerca MUR)
Record Dates: First submitted 2025-07-09; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: volounteers with different levels of social expertise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral and MR imaging (Experimental): After enrollment, participants will be screened on the basis of the inclusion and exclusion criteria. Subsequently, during the single study, participants will be administered a series of questionnaires (Edinburgh Handedness Inventory - Short Form; Evaluation of social related abilities, competences, and traits: Autism Quotient Test, DASS-21, SIAS, DERS, Ekman test; SET; I-TIPI, and conceptual ratings on semantic dimensions (moral, social, political). Then, an MR acquisition without contrast will be performed. Specifically, we will acquire structural, resting state and functional (BOLD) sequences, in the latter case during the administration of a semantic categorization task. The task is aimed to ascertain participants' responses time and accuracy in processing abstract concepts. Participants will be required to indicate the category of each of the visually presented words by means of button press. The study visit will last 3 hours in total.
  Interventions: Other: Behavioral and MR scanning

INTERVENTIONS:
Other: Behavioral and MR scanning — After enrollment, participants will be screened on the basis of the inclusion and exclusion criteria. Subsequently, during the single study, participants will be administered a series of questionnaires (Edinburgh Handedness Inventory - Short Form; Evaluation of social related abilities, competences, and traits: Autism Quotient Test, DASS-21, SIAS, DERS, Ekman test; SET; I-TIPI, and conceptual ratings on semantic dimensions (moral, social, political). Then, an MR acquisition without contrast will be performed. Specifically, we will acquire structural, resting state and functional (BOLD) sequences, in the latter case during the administration of a semantic categorization task. The task is aimed to ascertain participants' responses time and accuracy in processing abstract concepts. Participants will be required to indicate the category of each of the visually presented words by means of button press. The study visit will last 3 hours in total.

SUMMARY:
Social interaction is supported by several brain regions, which are involved in encoding socio-perceptual information, attributing affective and mental states to other conspecifics, and ultimately enabling the orchestration of an appropriate response. In this view, cognitive control mechanisms are necessary to select relevant information, allocate resources, and generate inferences. There is a close link between the mechanisms underlying social cognition and social conceptual knowledge, relating, for example, to abstract concepts such as "friendship". For example, children with autism spectrum disorder (ASD) show impairments in social interactions, and also in the ability to use all those abstract concepts that relate to internal states of the individual as well as to interactions between people.

Behavioral studies have shown how experience can impact the characterization of abstract concepts, influencing their personal, introspective, and contextual characteristics. Neuroimaging studies have also reported that, through mechanisms of brain plasticity, experience modulates neural networks shared with non-experts (e.g., by increasing brain volume and/or functional activity), but can also lead to the recruitment of additional brain resources, thus enriching the knowledge gained by experts. To date, the role of different types and levels of expertise in influencing the neural representation of specific categories of abstract concepts, and in particular social concepts, has not yet been fully elucidated.

DETAILED DESCRIPTION:
As human beings, we are embedded in social contexts, whether physical or virtual, that shape our brains throughout our lives, boosting our development, cognition and well-being. For us, interacting with others is an extremely simple thing, but it is actually one of the most complex computations our brains can perform. Indeed, when interacting with others, several regions of the brain are activated in order to encode socio-perceptual information, to attribute mental states to the interlocutors, and finally to trigger appropriate responses. Social interaction engages also by brain regions supporting social conceptual knowledge, relating, for example, to abstract concepts such as "friendship". Crucially, conceptual knowledge acquisition and organization are sustained by language. The mechanisms underlying social cognition and social conceptual knowledge are closely linked. This link relates, for example, to abstract concepts such as "friendship." For example, children with autism spectrum disorder (ASD) show impairments in social interactions and in the ability to use abstract concepts related to internal states of the individual as well as to interactions between people. Behavioral studies have shown how experience can impact the characterization of abstract concepts. This impact influences their personal, introspective, and contextual characteristics. Neuroimaging studies have also reported that experience modulates neural networks shared with non-experts. This happens through mechanisms of brain plasticity. Examples include increasing brain volume and/or functional activity. However, experience can also lead to the recruitment of additional brain resources. This enriches the knowledge gained by experts. Proficiency in a second language is another example of lifelong experience. Successful mastery of a second language requires the ability to switch between languages, inhibiting the unnecessary language and selecting the necessary one during interaction. Thus, second language proficiency modulates cognitive control functions and underlying neural structures and may influence social decision-making. The question of whether and how second language knowledge modulates the semantic control network is currently debated. The role of different types and levels of expertise in influencing the neural representation of specific categories of abstract concepts, particularly social concepts, has yet to be fully elucidated.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study
2. Male or female, aged between 25 and 50 years
3. Right-handed dominance
4. Normal vision or hypo-vision corrected with contact lenses
5. Participant must have different levels of social expertise, in order to be assigned to one of the following groups: (1) participants with subclinical social skills dysfunction, parents of children with Autism Spectrum Disorder, (2) participants with no specific social expertise, and (3) participants with high social expertise, namely social media influencers and politicians.

Exclusion Criteria:

1. Clinical and/or anamnestic evidence of neurological, psychiatric, or systemic disorders
2. Drug addiction and/or abuse of neuroactive drugs;
3. Contraindications and incompatibilities with MRI, and specifically presence of para-magnetic or ferro-magnetic metal body prostheses; presence of permanent biomedical implants (e.g., pacemakers, neuro-stimulators); pregnancy status; claustrophobia. Pregnancy status will be self-reported by the participants.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between participants' accuracy rate and BOLD signal | baseline
  Evaluate whether and how social expertise modulate the neural representation of different types of abstract concepts, and in particular social concepts.

SECONDARY OUTCOMES:
Correlation between participants' accuracy rate and scores in Autism Quotient Test, DASS-21, SIAS, DERS, Ekman test, SET and I-TIPI | baseline
  Evaluate whether and how individual affective and social characteristics modulate the characterization and the neural representation of different types of abstract concepts, and in particular social concepts.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Eccellenza Risonanza Magnetica ad Alto Campo (CERMAC), Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buchweitz A, Shinkareva SV, Mason RA, Mitchell TM, Just MA. Identifying bilingual semantic neural representations across languages. Brain Lang. 2012 Mar;120(3):282-9. doi: 10.1016/j.bandl.2011.09.003. Epub 2011 Oct 5. PMID 21978845
- [Background] Abutalebi J, Della Rosa PA, Ding G, Weekes B, Costa A, Green DW. Language proficiency modulates the engagement of cognitive control areas in multilinguals. Cortex. 2013 Mar;49(3):905-11. doi: 10.1016/j.cortex.2012.08.018. Epub 2012 Sep 1. PMID 23021069
- [Background] Del Maschio, N., Abutalebi, J., Schwieter, J., & Paradis, M. Language Organization in the Bilingual and Multilingual Brain. 2019 Feb; pp. 197-213. https://doi.org/10.1002/9781119387725.ch9
- [Background] Borghi AM, Binkofski F, Castelfranchi C, Cimatti F, Scorolli C, Tummolini L. The challenge of abstract concepts. Psychol Bull. 2017 Mar;143(3):263-292. doi: 10.1037/bul0000089. Epub 2017 Jan 16. PMID 28095000
- [Background] Bang J, Burns J, Nadig A. Brief report: Conveying subjective experience in conversation: production of mental state terms and personal narratives in individuals with high functioning autism. J Autism Dev Disord. 2013 Jul;43(7):1732-40. doi: 10.1007/s10803-012-1716-4. PMID 23179342
- [Background] Baez S, Garcia AM, Ibanez A. The Social Context Network Model in Psychiatric and Neurological Diseases. Curr Top Behav Neurosci. 2017;30:379-396. doi: 10.1007/7854_2016_443. PMID 27130326
- [Background] Conca F, Catricala E, Canini M, Petrini A, Vigliocco G, Cappa SF, Della Rosa PA. In search of different categories of abstract concepts: a fMRI adaptation study. Sci Rep. 2021 Nov 19;11(1):22587. doi: 10.1038/s41598-021-02013-8. PMID 34799624
- [Background] Binney RJ, Ramsey R. Social Semantics: The role of conceptual knowledge and cognitive control in a neurobiological model of the social brain. Neurosci Biobehav Rev. 2020 May;112:28-38. doi: 10.1016/j.neubiorev.2020.01.030. Epub 2020 Jan 23. PMID 31982602
- [Background] Adolphs R. Conceptual challenges and directions for social neuroscience. Neuron. 2010 Mar 25;65(6):752-67. doi: 10.1016/j.neuron.2010.03.006. PMID 20346753
- [Background] Wolf SM, Paradise J, Caga-anan C. The law of incidental findings in human subjects research: establishing researchers' duties. J Law Med Ethics. 2008 Summer;36(2):361-83, 214. doi: 10.1111/j.1748-720X.2008.00281.x. PMID 18547206